CLINICAL TRIAL: NCT01213225
Title: Geriatric Education and Its Effect on Certain Aspects of Hospital Care of the Nursing Home Patients - 12 Month Retrospective Study
Status: Completed | Type: Observational
Sponsor: Maimonides Medical Center (Other)
Responsible Party: Sergey Genkin, MD, Maimonides Medical Center
Other Study IDs: gerivsnot12month
Record Dates: First submitted 2010-09-29; First posted 2010-10-01 (Estimated); Last update posted 2011-08-18 (Estimated); Status verified 2011-08

CONDITIONS: Frail Elderly; Elderly; Hospitalization; Geriatrics
Keywords: Elderly; Hospitalization; Geriatrics; Mortality; Readmission; Length of Stay

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Nursing home patients admitted to the hospital poses significant challenge for health care providers. Geriatric teaching pays particular attention to these admissions and related problems. However, it yet to be proven, that geriatric training helps to overcome any of them in better way then non-geriatric education. The study aims to prove that geriatric care provides advantages over non-geriatric training in caring for nursing home patients admitted to the hospital.

DETAILED DESCRIPTION:
Context Nursing home patients admitted to the hospital poses significant challenge for health care providers. Geriatric age, frailty, multiple readmissions, prolonged length of stay, and high mortality are just few attributes of nursing home patients in the hospital. Geriatric teaching pays particular attention to these challenging problems. However, it yet to be proven, that geriatric training helps to overcome any of them in better way then non-geriatric education.

Objective To test the hypothesis that geriatric care provides advantages over non-geriatric training in caring for nursing home patients admitted to the hospital in regards to length of stay, rate of expirations and rate of readmissions. The secondary objective is to compare expirations and readmissions among patients cared for by geriatricians and non-geriatricians.

Design, Setting, and Participants Retrospective cohort study of patients admitted from Metropolitan Jewish Geriatric Nursing Home (MJGNH) to Maimonides Medical Center (MMC) over 12 month period and under the care of geriatricians, non-geriatric internists, and surgeons. Comparison of the three study groups by age, sex, expiration rate, length of hospital stay (LOS) and readmission rate. Comparison of expired patients by age, sex and average LOS. Comparison of readmissions expiration rate, by preservation of continuity of care, by emergency room visits without admission.

ELIGIBILITY:
Inclusion Criteria:

* all patients admitted to Maimonides Medical Center (MMC) from affiliated Metropolitan Jewish Geriatric Nursing Home (MJGNH)for '12 month period.

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 65 years of age and older
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2010-12

CONTACTS AND LOCATIONS:
Overall Officials: Sergey I Genkin, Principal Investigator — Maimonides Medical Center